CLINICAL TRIAL: NCT04719715
Title: Evaluation of ANCA Testing by Antigen Specific Assays in Small Vessel Vasculitis
Brief Title: Evaluation of Anti-neutrophil Cytoplasm Antibodies Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mai Mahmoud Fahmy Mansour, Assistant lecturer of Rheumatology, Rehabilitation and Physical Medicine, Sohag University
Other Study IDs: ANCA testing evaluation
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Immunological Testing in Small-vessel Vasculitis
Keywords: ANCA vasculitis, ANCA testing, antigen specific essays, IIF
MeSH Terms: interventions — Fluorescent Antibody Technique, Indirect

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with ANCA vasculitis: Indirect immunofluorescence (IIF) will be performed as well as myeloperoxidase antibody(MPO)- and anti-proteinase 3 (PR3-) ANCA immunoassays and evaluated
  Interventions: Diagnostic Test: Indirect immunofluorescence (IIF) , myeloperoxidase antibody(MPO)- and anti-proteinase 3 (PR3-) ANCA immunoassays
- Controls with autoimmune diseases other than ANCA vasculitis: Indirect immunofluorescence (IIF) will be performed as well as myeloperoxidase antibody(MPO)- and anti-proteinase 3 (PR3-) ANCA immunoassays and evaluated
  Interventions: Diagnostic Test: Indirect immunofluorescence (IIF) , myeloperoxidase antibody(MPO)- and anti-proteinase 3 (PR3-) ANCA immunoassays

INTERVENTIONS:
Diagnostic Test: Indirect immunofluorescence (IIF) , myeloperoxidase antibody(MPO)- and anti-proteinase 3 (PR3-) ANCA immunoassays — Measurement and evaluation of the ANCA testing

SUMMARY:
Anti-neutrophil cytoplasm antibodies (ANCA) are defined as important serological markers for the diagnosis of some forms of small vessel vasculitis, including granulomatosis with polyangiitis (GPA) , microscopic polyangiitis(MPA) and to a lesser extent Churg -Strauss syndrome or Eosinophilic granulomatosis with polyangiitis (EGPA).So they are called ANCA-associated vasculitis(AAV).

An international consensus statement for ANCA testing statement was issued in 2017 and states that the antigen specific immunoassays can be used for the accurate diagnosis of ANCA-associated vasculitis without the need for indirect immunofluorescence(IIF). In the present study we will test whether the antigen specific assays screening is a valuable alternative to IIF confirming with immunoassay for the diagnosis of AAV on a number of patients and controls.

Aim To evaluate the performance of the recommended strategy for the detection of ANCA based on screening with antigen specific immunoassays on a number of AAV patients and relevant disease controls In Kagawa university hospital (rheumatology department).

Patients and methods This is a prospective study will be conducted at the department of rheumatology in Kagawa university hospital in which consecutive samples will be included from patients suspected to have AAV; patients subsequently identified as having AAV will be included as AAV patients, while patients in which the diagnosis AAV is rejected, will be included as disease controls. PR3-and MPO-ANCA will be performed using assays from Medical & Biological Laboratories Co (Anchor CLEIA) isayama.takuya@mbl.co.jp

DETAILED DESCRIPTION:
To evaluate the performance of the recommended strategy for the detection of ANCA based on screening with antigen specific immunoassays on a number of AAV patients and relevant disease controls (i. e., patients for whom ANCA would be requested in the context of small-vessel vasculitis such as patients with infections, drug-induced diseases, connective tissue disease, etc.).

ELIGIBILITY:
Inclusion Criteria:

.All patients included must be older than 18 years and able to give informed consent.

* Classification criteria and nomenclature for AAV are from the American College of Rheumatology
* Serum sampling should be done before initiation of immunosuppressive treatment or no later than 2 weeks after onset of low-medium dose of immunosuppressive treatment (but this should be documented)

Exclusion Criteria:

.Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Anti-proteinase 3 antibody (PR3), anti-myeloperoxidase (MPO) antibody presence in patients with small-vessel vasculitis versus patients without vasculitis | within two weeks of immunosuppressive treatment not after that
  Antibodies are detected using chemiluminescent enzyme immunoassay (CLEIA).Values above 3.5 u/ml are considered positive

CONTACTS AND LOCATIONS:
Overall Officials: Mai Mansour, Principal Investigator — Sohag University
Locations (1):
- Kagawa univeristy, Hiragi, Kagawa-ken, Japan

IPD SHARING:
Plan to Share IPD: No